CLINICAL TRIAL: NCT02373462
Title: Effect of olmesaRtan on Walking distancE and quaLIty of lifE in Peripheral Artery Disease Patients With Hypertension Treated For Intermittent Claudication (RELIEF)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The data of the paper referenced in the preparation of the protocols in this task were manipulated and the paper was withdrawn.
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2014-0888
Record Dates: First submitted 2015-02-14; First posted 2015-02-27 (Estimated); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Peripheral Artery Disease With Intermittent Claudication
MeSH Terms: interventions — olmesartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- olmesartan group (Experimental): olmesartan (20mg qd then 40mg qd for titrating BP <140/90 mmHg)
  Interventions: Drug: Olmesartan
- other group (Active Comparator): other anti-hypertensive drug (titrating BP <140/90 mmHg)
  Interventions: Drug: other anti-hypertensive drug

INTERVENTIONS:
Drug: Olmesartan
  Arms: olmesartan group
Drug: other anti-hypertensive drug — CCB, diuretics, alpha blocker, direct vasodilator, beta blocker
  Arms: other group

SUMMARY:
To study the effect of olmesartan on walking distance and quality of life in peripheral artery disease patients with hypertension treated For intermittent claudication.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20 and 85 years at visit 1
* Patients with ankle-brachial index (ABI) of less than 0.9 in one or both legs with history of intermittent claudication stable for the previous 6 months
* Patients whose statins, anti hypertensive medications and antiplatelet medications are stable for the past 6 months. Statins and cilostazol are allowed but needs to be stable for the past 6 months (diabetic medications may be changed)
* Patients whose blood pressure is more than 140/90 mmHg with/without anti-hypertension treatment

Exclusion Criteria:

* Blood pressure of more than 180/110 mmHg
* Patients taking ARBs or ACE inhibitors treatment for at least 6 months before
* Patients taking aldosterone receptor antagonists at least 6 months before
* Patients with serum creatinine of more than 3 mg/dL
* serum potassium (K+) > 5.5mg/dl
* History of bilateral renal artery stenosis
* History of acute coronary syndrome or heart failure hospitalization within 6 months
* Peripheral arterial revascularization planned within 1 month
* Critical limb ischemia
* Patients with impaired cognition (e.g. dementia)
* pregnancy or women at age of childbearing potential

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-08-25 (Actual); Primary Completion 2015-11-17 (Actual); Study Completion 2015-11-17 (Actual)

PRIMARY OUTCOMES:
Pain free maximum walking distance and time | 12th week
  Effect of olmesartan in maximum, pain free walking distance & time

SECONDARY OUTCOMES:
Quality of life as measured by questionnaires | 24th week
  Effect of olmesartan in quality of life (WIQ, SF-36)

OTHER OUTCOMES:
Pulse wave analysis as measured by PWV | 24th week
  pulse wave velocity
Blood pressure by measured by 24hr ABPM | 24th week
  24hr ambulatory blood pressure monitoring

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Department of Internal Medicine, Severance Hospital, Seoul, South Korea